CLINICAL TRIAL: NCT06569732
Title: Clinical Efficacy, Feasibility, and Cost-effectiveness of Homemade Oral Nutrition Supplements on Patients on Hemodialysis With Protein-energy Wasting: a Parallel, Open-labeled, Randomized Controlled Trial
Brief Title: Effects of Homemade Oral Nutrition Supplements for Patients on Hemodialysis With Protein-energy Wasting
Acronym: HOMES-HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Malaysia Sabah (Other)
Collaborators: National Kidney Foundation Malaysia (Unknown)
Responsible Party: Principal Investigator, Khor Ban Hock, Senior Lecturer, Universiti Malaysia Sabah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS2409
Record Dates: First submitted 2024-07-28; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Protein-Energy Wasting; Kidney Failure; Hemodialysis
Keywords: hemodialysis; protein-energy wasting; kidney failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homemade oral nutrition supplements (Experimental): Homemade oral nutrition supplements, 200 ml/day
  Interventions: Other: Homemade oral nutrition supplements
- Commercial oral nutrition supplements (Active Comparator): Commercial oral nutrition supplements, 200 ml/day
  Interventions: Other: Commercial oral nutrition supplements

INTERVENTIONS:
Other: Homemade oral nutrition supplements — The homemade oral nutrition supplement is made of soy milk, whey protein powder, vegetable oil, and fruit juices
  Arms: Homemade oral nutrition supplements
Other: Commercial oral nutrition supplements — The commercial oral nutrition supplement is kidney-specific oral nutrition supplement that is high in energy and protein, but low in electrolytes and fluid
  Arms: Commercial oral nutrition supplements

SUMMARY:
The goal of this clinical trial is to learn if homemade oral nutrition supplements works to treat protein energy wasting in patients on hemodialysis. It will also learn about the cost-effectiveness of homemade oral nutrition supplements. The main questions it aims to answer are:

* Does homemade oral nutrition supplements improve the nutritional status of patients on hemodialysis with protein energy wasting?
* What is the cost-effectiveness of homemade oral nutrition supplements?

Researchers will compare homemade oral nutrition supplements to commercial oral nutrition supplements to see if homemade oral nutrition supplements works to treat protein energy wasting in patients on hemodialysis.

Participants will:

* Take homemade or commercial oral nutrition supplements every day for 6 months
* Have assessment of nutritional status performed by researchers every three monthly

ELIGIBILITY:
Inclusion Criteria:

* on maintenance HD dialysis treatment (thrice weekly and 4-hour per session) for at least three months
* age 18 - 70 year old
* diagnosed with protein energy wasting using the malnutrition inflammation score (≥ 5)

Exclusion Criteria:

* a history of poor adherence to HD treatment (frequently miss the HD treatment for more than one session every month)
* a history of frequent hospitalization (more than once in the past one month)
* on regular oral nutrition supplements
* diagnosed with malignancy
* pregnant or lactating women
* allergic to study products such as soy milk or milk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Malnutrition Inflammation Score at 3-month and 6-month | Baseline, 3-month, and 6-month
  The Malnutrition Inflammation Score is a composite score used to determine protein energy wasting. It consists of 10 questions, each rated on a scale from 0 to 3. The total score ranges from 0 to 30, with higher scores indicating more severe malnutrition and inflammation. A score of 5 or above suggests the presence of protein-energy wasting.

SECONDARY OUTCOMES:
Changes from baseline in skeletal muscle mass at 3-month and 6-month | Baseline, 3-month, and 6-month
  The skeletal muscle mass will be measured using a bio-impedance spectroscopy ro determine muscle mass and fat mass
Changes from baseline in body fat mass at 3-month and 6-month | Baseline, 3-month, and 6-month
  The body fat mass will be measured using a bio-impedance spectroscopy ro determine muscle mass and fat mass
Changes from baseline in energy intake at 3-month and 6-month | Baseline, 3-month, and 6-month
  The energy intake will be assessed using 24-hour diet recall forms
Changes from baseline in protein intake at 3-month and 6-month | Baseline, 3-month, and 6-month
  The protein intake will be assessed using 24-hour diet recall forms
Changes from baseline in intradialytic weight change at 3-month and 6-month | Baseline, 3-month, and 6-month
  The intradialytic weight change will be determined based on difference in post-dialysis and pre-dialysis weight of the next dialysis session
Changes from baseline in serum albumin at 3-month and 6-month | Baseline, 3-month, and 6-month
  Serum albumin will be obtained from the participants' routine blood test
Changes from baseline in serum phosphorus at 3-month and 6-month | Baseline, 3-month, and 6-month
  Serum phosphorus will be obtained from the participants' routine blood test
Changes from baseline in serum potassium at 3-month and 6-month | Baseline, 3-month, and 6-month
  Serum potassium will be obtained from the participants' routine blood test
Changes from baseline in handgrip strength at 3-month and 6-month | Baseline, 3-month, and 6-month
  Handgrip strength will be measured using a digital hand dynamometer
Cost-Effectiveness Ratio | 6-month
  The cost-effectiveness ratio will be calculated by dividing the cost of oral nutrition supplements (unit in Malaysia ringgit) for 6 months with the change in malnutrition inflammation score from baseline to 6-month (refer primary outcome 1). In this analysis, there is no minimum or maximum values, but a lower value indicates better cost-effectiveness (lower cost with a greater health benefit).
Acceptability of oral nutrition supplements | 6-month
  A questionnaire will be used to assess product acceptance using a 5-point Likert scale. The scale ranges from 1 to 5, with higher scores indicating greater acceptance of the product. The questionnaire consists of 5 questions, so the total score ranges from a minimum of 5 to a maximum of 25.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Hock Khor, PhD, Principal Investigator — Universiti Malaysia Sabah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahathevan S, Karupaiah T, Khor BH, Sadu Singh BK, Mat Daud ZA, Fiaccadori E, Sabatino A, Chinna K, Abdul Gafor AH, Bavanandan S, Visvanathan R, Yahya R, Wahab Z, Goh BL, Morad Z, Bee BC, Wong HS. Muscle Status Response to Oral Nutritional Supplementation in Hemodialysis Patients With Protein Energy Wasting: A Multi-Center Randomized, Open Label-Controlled Trial. Front Nutr. 2021 Dec 10;8:743324. doi: 10.3389/fnut.2021.743324. eCollection 2021. PMID 34977109
- [Background] Sahathevan S, Khor BH, Ng HM, Gafor AHA, Mat Daud ZA, Mafra D, Karupaiah T. Understanding Development of Malnutrition in Hemodialysis Patients: A Narrative Review. Nutrients. 2020 Oct 15;12(10):3147. doi: 10.3390/nu12103147. PMID 33076282